CLINICAL TRIAL: NCT02744755
Title: A Randomized, Double-blind, Parallel-group, Multicenter Study to Demonstrate Similar Efficacy and to Compare Safety and Immunogenicity of GP2017 and Humira® in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: Clinical Trial to Compare Treatment With GP2017 and Humira® in Patients With Rheumatoid Arthritis
Acronym: ADMYRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Collaborators: Hexal AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GP17-302; 2015-003433-10 (EudraCT Number)
Record Dates: First submitted 2016-04-12; First posted 2016-04-20 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GP2017

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GP2017 (Experimental): Group 1 will receive treatment with 40mg GP2017 (Adalimumab - GP2017) by subcutaneous injection every other week up to 24 weeks (Study Period 1) at which patients achieving at least a moderate clinical response continue treatment with 40mg GP2017 subcutaneous injection every other week up to 48 weeks (Study Period 2).
  Interventions: Biological: Adalimumab - GP2017
- US Licensed Humira (Active Comparator): Group 2 will receive treatment with 40mg Humira® (Adalimumab - US licensed Humira®) by subcutaneous injection every other week up to 24 weeks (Study Period 1) at which patients achieving at least a moderate clinical response will be switched to treatment with 40mg GP2017 subcutaneous injection every other week up to 48 weeks (Study Period 2).
  Interventions: Biological: Adalimumab - US licensed Humira

INTERVENTIONS:
Biological: Adalimumab - GP2017 — Adalimumab - GP2017
  Other Names: GP2017
  Arms: GP2017
Biological: Adalimumab - US licensed Humira — Adalimumab - US licensed Humira
  Other Names: Humira - Comparator
  Arms: US Licensed Humira

SUMMARY:
Clinical trial to compare treatment with GP2017 and Humira® in patients with Rheumatoid Arthritis

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate similar efficacy and safety of GP2017 and US-licensed Humira® in patients with moderate to severe rheumatoid arthritis (RA) with inadequate response to Disease modifying anti-rheumatic drugs (DMARDs), including methotrexate (MTX).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have been diagnosed with RA ≥ 6 months prior to screening
2. Patients must have active disease, defined as DAS28-CRP ≥ 3.2 at the time of screening
3. Patients must have CRP levels above 5mg/l or ESR levels above the upper limits of normal
4. Patients must have had inadequate clinical response to MTX 10 - 25 mg/week

Exclusion Criteria:

1. Previous treatment with adalimumab, other anti-TNFα therapies or cell depleting agents, e.g. anti-CD20 therapy
2. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during treatment
3. Nursing (lactating) or pregnant women
4. History of or ongoing inflammatory or autoimmune diseases other than RA, e.g. mixed connective tissue disease, systemic lupus erythematosus etc.
5. Systemic corticosteroids > 7.5mg/day within 4 weeks prior to baseline
6. History or presence of cancer or lymphoproliferative disease other than a successfully and completely treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix and/or removed non-invasive colon polyps, with no evidence of recurrence
7. History of uncontrolled diabetes, unstable ischemic heart disease, congestive heart failure (New York Heart Association III-IV), active peptic ulcer disease, recent stroke (within 3 months)
8. Subject known to have immune deficiency, history of positive human immunodeficiency virus (HIV) status or immunocompromised for other reasons
9. History of clinically significant hematologic (e.g. severe anemia, leucopenia, thrombocytopenia), renal or liver disease (e.g. glomerulonephritis, fibrosis, cirrhosis, hepatitis)
10. History of persistent chronic infection; recurrent infection or active infections
11. History of tuberculosis, presence of active tuberculosis, latent tuberculosis as detected by imaging (e.g. chest X-ray, chest Computerized Tomography(CT) scan, Magnetic Resonance Imaging (MRI)) and/ or positive QuantiFERON-TB Gold test (QFT)
12. History or evidence of opportunistic infections, e.g. histoplasmosis, listeriosis, legionellosis
13. Positive serology Hepatitis B (either HBsAg or anti-HBc) or Hepatitis C (positive HCV-Ab or HCV-RNA) indicative of previous or current infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (83):
- United States (30):
  - Arizona Arthritis & Rheumatology, Mesa, Arizona
  - Sun Valley Arthritis Center Ltd., Peoria, Arizona
  - Medvin Clinical Research, Covina, California
  - MD Med Corp, Hemet, California
  - Talbert Medical Group, Huntington Beach, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Joao Nascimento (Private Practice), Bridgeport, Connecticut
  - Arthritis & Rheumatic Disease Specialties, Aventura, Florida
  - RASF - Clinical Research Center, Boca Raton, Florida
  - QPS MRA (Miami Research Associates), Miami, Florida
  - Omega Research Consultants Orlando, Orlando, Florida
  - Family Clinical Trials, LLC., Pembroke Pines, Florida
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - McIlwain Medical Group, PA, Tampa, Florida
  - BayCare Medical Group, Inc, Tampa, Florida
  - Lovelace Scientific Resources, Inc., Venice, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Marietta Rheumatology Associates, PC, Marietta, Georgia
  - Center for Arthritis & Osteoporosis, Elizabethtown, Kentucky
  - Arthritis and Rheumatology Consultants, Edina, Minnesota
  - Physician Research Collaboration, Lincoln, Nebraska
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Montefiore Medical Center PRIME, Lake Success, New York
  - Medication Management, LLC, Greensboro, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Low Country Rheumatology, PA, North Charleston, South Carolina
  - Ramesh C Gupta, MD, Memphis, Tennessee
  - Austin Regional Clinic, P.A., Austin, Texas
  - Tekton Research, Inc., Austin, Texas
  - Sentara Medical Group Clinical Research, Norfolk, Virginia
- Czechia (5):
  - IMEDICA s.r.o., Brno
  - Revmacentrum MUDr. Mostera s.r.o., Brno-Židenice
  - Revmatologicka a interni ambulance, Kladno
  - Revmatologicky Ustav, Prague
  - MEDICAL PLUS s.r.o., Uherské Hradiště
- Germany (3):
  - Praxis Dr. Walter, Rendsburg, Schleswig-Holstein
  - Rheumatologische Schwerpunktpraxis Steglitz, Berlin
  - HRF Hamburger Rheuma Forschungszentrum, Hamburg
- Hungary (6):
  - Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaz, Békéscsaba
  - Sopron Medical Egeszsegugyi Szolgaltato Kft., Budapest
  - Hevizgyogyfurdo es Szent Andras Reumakorhaz Reumatologia III, Hévíz
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz Reumatologiai Osztaly, Nyíregyháza
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Vital Medical Center, Veszprém
- Italy (2):
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan
  - A.O.U. Senese Policlinico Santa Maria alle Scotte UOC Reumatologia, Siena
- Malaysia (5):
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Sibu, Sibu, Sarawak
  - Hospital Selayang, Batu Caves, Selangor
- Mexico (6):
  - Centro Investigacion en Artritis y Osteoporosis S.C., Mexicali, Baja California Norte
  - Centro de Alta Especialidad en Reumatología e Investigación del Potosí, S.C., San Luis Potosí City, San Luis Potos
  - Clinical Research Institute S.C., Tlalnepantla, State of Mexico
  - Investigacion y Biomedicina de Chihuahua, S.C., Chihuahua City
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - RM Pharma Specialists SA de CV, México
- Poland (8):
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela Dept of Clinical Reumatology, Bydgoszcz
  - Centrum Kliniczno - Badawcze J. Brzezicki, B. Górnikiewicz-Brzezicka Lekarze Spółka Partnerska, Elblag
  - Centrum Medyczne Pratia Gdynia ProFamilia Spolka Akcyjna, Oddzial w Gdyni, Gdynia
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska sp. komandytowo-akcyjna, Lodz
  - Ai Centrum Medyczne Sp. Z O.O. Sp.K., Poznan
  - RCMed, Sochaczew
  - Slaskie Centrum Reumatologii,Rehabilitacji i Zapobiegania Niepelnosprawnosci im. Gen. Jerzego Zietka, Ustroń
  - Niepubliczny Zakład Opieki Zdrowotnej "Biogenes" Sp. z o.o., Wroclaw
- Romania (5):
  - Spitalul Clinic Judetean de Urgenta Brasov Sectia Reumatologie, Brasov
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca Sectia Reumatologie, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta "Sf. Apostol Andrei" Galati Sectia Reumatologie, Galati
  - RK Medcenter SRL, Iași
  - Spitalul Municipal Ploiesti Sectia Reumatologie, Ploieşti
- Russia (5):
  - SBIH of Nizhniy Novgorod region " City Clinical Hospital # 5", Nizhny Novgorod
  - SPb SBIH "Clinical Rheumatological Hospital # 25", Saint Petersburg
  - Research Institute of Emergency Medical Care, Saint Petersburg
  - SHI Ulyanovsk Reg Clinical Hospital, Ulyanovsk
  - SBHI of Yaroslavl Region "Clinical Hospital #3", Yaroslavl
- Serbia (2):
  - Institute of Rheumatology, Belgrade
  - Special Hospital for Rheumatic Diseases, Novi Sad
- Spain (4):
  - Hospital de Cruces, Barakaldo
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Infanta Luisa, Seville
- United Kingdom (2):
  - Princess Alexandra Hospital; Dept of Rheumatology; Williams Day Unit, Harlow, Essex
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blauvelt A, Leonardi CL, Gaylis N, Jauch-Lembach J, Balfour A, Lemke L, Hachaichi S, Brueckmann I, Festini T, Wiland P. Treatment with SDZ-ADL, an Adalimumab Biosimilar, in Patients with Rheumatoid Arthritis, Psoriasis, or Psoriatic Arthritis: Results of Patient-Reported Outcome Measures from Two Phase III Studies (ADMYRA and ADACCESS). BioDrugs. 2021 Mar;35(2):229-238. doi: 10.1007/s40259-021-00470-1. Epub 2021 Mar 2. PMID 33651341
- [Derived] Huizinga TWJ, Torii Y, Muniz R. Adalimumab Biosimilars in the Treatment of Rheumatoid Arthritis: A Systematic Review of the Evidence for Biosimilarity. Rheumatol Ther. 2021 Mar;8(1):41-61. doi: 10.1007/s40744-020-00259-8. Epub 2020 Dec 1. PMID 33263165
- [Derived] Wiland P, Jeka S, Dokoupilova E, Brandt-Jurgens J, Miranda Limon JM, Cantalejo Moreira M, Cabello RV, Jauch-Lembach J, Thakur A, Haliduola H, Brueckmann I, Gaylis NB. Switching to Biosimilar SDZ-ADL in Patients with Moderate-to-Severe Active Rheumatoid Arthritis: 48-Week Efficacy, Safety and Immunogenicity Results From the Phase III, Randomized, Double-Blind ADMYRA Study. BioDrugs. 2020 Dec;34(6):809-823. doi: 10.1007/s40259-020-00447-6. PMID 33119861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 353 patients were randomized (1:1)and received at least one dose of study drug; 303 patients completed the study.Eligible patients in the Humira group who completed Study Period 1 (baseline to week 24) with an at least moderate response by DAS28-CRP score were switched to GP2017 treatment during Study Period 2 (Week 24 to week 48).
Pre-assignment Details: Full analysis set: randomized patients (study drug assigned) Per protocol set study period 1 (SP1) / study period 2(SP2): patients who completed Week 12 (SP1) / Week 48 (SP2) without major protocol deviations and received at least 5 doses of study drug up to Week 10 (SP1) / 10 doses of IMP from Week 24 to Week 46 (SP2)
Groups:
- GP2017: Group 1 received treatment with 40 mg GP2017 in 0.8 mL of solution administered subcutaneously from pre-filled syringes up to 24 weeks (study Period 1) after which patients achieving at least a moderate clinical response continued treatment with 40mg GP2017 subcutaneous injection up to 46 weeks (study Period 2).
- Humira / Switched GP2017: Group 2 received treatment with 40 mg Humira in 0.8 mL of solution administered subcutaneously from pre-filled syringes up to 24 weeks (study Period 1) after which patients achieving at least a moderate clinical response were switched to 40mg GP2017 subcutaneous injection up to 46 weeks (study Period 2).
Period: Study Period 1
Arm/Group | GP2017 | Humira / Switched GP2017
Started (randomized) | 177 | 176
Completed (completed study period 1) | 163 | 168
Not Completed | 14 | 8
Not completed — Protocol Violation | 2 | 1
Not completed — not defined | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 8 | 4
Period: Study Period 2
Arm/Group | GP2017 | Humira / Switched GP2017
Started | 159 | 166
Completed | 145 | 158
Not Completed | 14 | 8
Not completed — Adverse Event | 5 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — not defined | 3 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lack of Efficacy | 3 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for Study Period 1 Full Analysis Set (SP 1 FAS ). The SP 1 FAS is comprised of all randomized patients to whom study treatment has been assigned.
Groups:
- Total: Total of all reporting groups
Arm/Group | GP2017 | Humira / Switched GP2017 | Total
Number analyzed (Participants) | 177 | 176 | 353
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline characteristics are presented for Study Period 1 Full Analysis Set (SP 1 FAS ). The SP 1 FAS is comprised of all randomized patients to whom study treatment has been assigned.
  years | 52.8 (12.81) | 53.8 (12.22) | 53.3 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics are presented for Study Period 1 Full Analysis Set (SP 1 FAS ). The SP 1 FAS is comprised of all randomized patients to whom study treatment has been assigned.
  Participants
    Female | 153 | 142 | 295
    Male | 24 | 34 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics are presented for Study Period 1 Full Analysis Set (SP 1 FAS ). The SP 1 FAS is comprised of all randomized patients to whom study treatment has been assigned.
  Participants
    White | 152 | 152 | 304
    American Indian or Alaska Native | 14 | 15 | 29
    Black or African American | 6 | 3 | 9
    Asian | 1 | 3 | 4
    Other | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Study Period 1: Change in DAS28-CRP Score From Baseline at Week 12 in Patients Treated With GP2017 and Patients Treated With Humira
Description: Disease activity score (DAS) 28-CRP is based on 28-joint count (tender and swollen joints), C-reactive protein and patient's assessment of global disease activity (GDA) or general health (GH), values range from 0.96 to 10.0 while higher values mean a higher disease activity. • A DAS28-CRP value >5.1 corresponds to a high disease activity • A DAS28-CRP value between 3.2 and 5.1 corresponds to a moderate disease activity • A DAS28-CRP value between 2.6 and 3.2 corresponds to a low disease activity • A DAS28-CRP value < 2.6 corresponds to remission DAS28-CRP = 0.56 * sqrt(tender28) + 0.28* sqrt(swollen28) + 0.36 * ln(CRP+1) + 0.014 * GDA or GH + 0.96 where • tender28 and swollen28 are the number of tender and swollen joints as assessed using 28-joint count • CRP is C-reactive protein (mg/l) • GDA is the global disease activity measured on a Visual Analogue Scale (VAS) of 100 mm
Time Frame: Study period 1: week 12
Population: Treatment Period 1 Per-Protocol set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 140 | 144
scores on a scale | -2.16 (0.114) | -2.18 (0.110)
Statistical Analysis 1: Comparison: GP2017 vs Humira / Switched GP2017; Therapeutic equivalence in terms of change from baseline in DAS28-CRP at week 12 will be concluded if the 95% confidence interval for the LS mean difference between GP2017 and Humira is contained within the interval [-0.6; 0.6]. A mixed-model repeated measures analysis was performed for DAS28-CRP change from baseline including treatment, stratification factors, time, the interaction between time (visits) and treatment all as categorical variables, and baseline DAS28-CRP as a continuous variable; Test type: Equivalence — A 0.6 change in DAS28-CRP score is considered as no clinically meaningful difference by EULAR criteria and is therefore used as the equivalence margin limits [0.6,-0.6]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.24 to 0.27], Standard Error of Mean 0.129
Statistical Analysis 2: Comparison: GP2017 vs Humira / Switched GP2017; Therapeutic equivalence in terms of change from baseline in DAS28-CRP at week 12 will be concluded if the 90% confidence interval for the LS mean difference between GP2017 and Humira is contained within the interval [-0.6; 0.6]. A mixed-model repeated measures analysis was performed for DAS28-CRP change from baseline including treatment, stratification factors, time, the interaction between time (visits) and treatment all as categorical variables, and baseline DAS28-CRP as a continuous variable; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.02, 90% CI 2-sided [-0.19 to 0.23], Standard Error of Mean 0.129

2. Secondary Outcome: Study Period 1: Time-weighted Averaged Change From Baseline in DAS28-CRP Until Week 24 in Patients Treated With GP2017 and With Humira
Description: as for outcome 1
Time Frame: Study period 1: week 24
Population: Treatment Period 1 Per-Protocol set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 127 | 138
scores on a scale | -1.85 (0.098) | -1.93 (0.092)
Statistical Analysis 1: Comparison: GP2017 vs Humira / Switched GP2017; ANCOVA model included treatment, body weight as per CRF, prior therapy as per CRF, region as per CRF as fixed effects and baseline DAS28-CRP values as covariate; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.11 to 0.27], Standard Error of Mean 0.096
Statistical Analysis 2: Comparison: GP2017 vs Humira / Switched GP2017; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Mean Difference (Final Values) = 0.08, 90% CI 2-sided [-0.08 to 0.24], Standard Error of Mean 0.096

3. Secondary Outcome: Study Period 1- Proportion of Patients Achieving EULAR Criterion for Remission
Description: Proportion of patients achieving European League against Rheumatism (EULAR) remission (defined as DAS28 CRP < 2.6 )
Time Frame: week 4, week 12 and week 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 127 | 138
Participants
  EULAR remission week 4: number analyzed (Participants) | 123 | 138
  EULAR remission week 4 | 15 | 7
  EULAR remission week 12: number analyzed (Participants) | 126 | 138
  EULAR remission week 12 | 32 | 38
  EULAR remission week 24 | 49 | 71

4. Secondary Outcome: Study Period 1- Proportion of Patients Achieving EULAR Criterion for Good Response
Description: Proportion of patients achieving European League against Rheumatism (EULAR) good response (defined as DAS28<=3.2 at post-baseline assessment timepoint(s) with an improvement of >1.2 in DAS28 from baseline.)
Time Frame: week 4, week 12 and week 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 127 | 138
Participants
  Good response week 4: number analyzed (Participants) | 123 | 138
  Good response week 4 | 22 | 25
  Good response week 12: number analyzed (Participants) | 126 | 138
  Good response week 12 | 51 | 63
  Good response week 24: number analyzed (Participants) | 126 | 138
  Good response week 24 | 76 | 93

5. Secondary Outcome: Study Period 1- Proportion of Patients Achieving EULAR Criterion for Moderate Response
Description: Proportion of patients achieving European League against Rheumatism (EULAR) moderate response (defined as DAS28<=3.2 at post-baseline assessment timepoint(s) with an improvement of >0.6 to <=1.2 from baseline or DAS28 >3.2 to <=5.1 with an improvement of >0.6 to <=1.2 or of >1.2 from baseline or DAS28 >5.1 with an improvement of >1.2 from baseline) ;
Time Frame: week 4, week 12 and week 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 127 | 138
Participants
  Moderate response week 4: number analyzed (Participants) | 123 | 138
  Moderate response week 4 | 63 | 78
  Moderate response week 12: number analyzed (Participants) | 126 | 138
  Moderate response week 12 | 64 | 62
  Moderate response week 24: number analyzed (Participants) | 126 | 138
  Moderate response week 24 | 42 | 42

6. Secondary Outcome: Study Period 1- Proportion of Patients Achieving EULAR/ACR Boolean Remission Criteria
Description: Proportion of patients achieving EULAR/American College of Rheumatology (EULAR/ACR) Boolean remission criteria (defined as number of tender joint count 28 <=1 and swollen joint count 28 <=1, CRP level (mg/dL) <=1 and patient's global assessment <=1 on a scale of 1-10 (corresponding to <=10 on a scale of 1-100).
Time Frame: week 4, week 12, week 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 127 | 138
Participants
  week 4: number analyzed (Participants) | 123 | 138
  week 4 | 4 | 0
  week 12: number analyzed (Participants) | 126 | 138
  week 12 | 8 | 12
  week 24 | 19 | 26

7. Secondary Outcome: Study Period 1: Change in DAS28-CRP and DAS28-ESR Scores From Baseline to Week 24 in Patients Treated With GP2017 and Patients Treated With Humira
Description: DAS28-CRP is a disease activity score and defined in primary outcome measure. DAS28-ESR is the DAS28 erythrocyte sedimentation rate score.
  DAS28-CRP and DAS28-ESR:
  1. best is 0,
  2. < 2.6 - remission,
  3. ≥ 2.6 to ≤ 3.2 - low disease activity
  4. > 3.2 to ≤ 5.1 - moderate disease activity
  5. > 5.1 - high disease activity
  DAS28-ESR = 0.56 * sqrt(tender28) + 0.28*sqrt(swollen28) + 0.7 * ln(ESR) + 0.014 * GDA where • tender28 and swollen28 are the number of tender and swollen joints as assessed using 28-joint count • CRP is C-reactive protein (mg/l) • ESR is erythrocyte sedimentation rate (mm/h) • GDA is the global disease activity measured on a Visual Analogue Scale (VAS) of 100 mm.Values range from 0 to 10. Higher values mean a higher disease activity.
Time Frame: study period 1: week 2, 4, 24
Population: Treatment Period 1 Per-Protocol set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 127 | 138
scores on a scale
  DAS28 CRP week 2: number analyzed (Participants) | 122 | 137
  DAS28 CRP week 2 | -0.86 (0.107) | -0.92 (0.101)
  DAS28 CRP week 4: number analyzed (Participants) | 123 | 138
  DAS28 CRP week 4 | -1.31 (0.112) | -1.36 (0.105)
  DAS28 CRP week 24 | -2.61 (0.109) | -2.83 (0.103)
  DAS28 ESR week 2: number analyzed (Participants) | 125 | 137
  DAS28 ESR week 2 | -0.94 (0.115) | -0.98 (0.109)
  DAS28 ESR week 4: number analyzed (Participants) | 125 | 138
  DAS28 ESR week 4 | -1.51 (0.124) | -1.51 (0.117)
  DAS28 ESR week 24: number analyzed (Participants) | 126 | 138
  DAS28 ESR week 24 | -2.97 (0.127) | -3.16 (0.120)

8. Secondary Outcome: Study Period 1- Proportion of Patients Achieving ACR20/50/70 Response at Weeks 4, 12 and 24
Description: ACR20 response was defined if a patient fulfilled all 3 criteria below: -at least 20% improvement in tender 68 joint count
  -at least 20% improvement in swollen 66 joint-count; And at least 20% improvement in at least 3 of the following 5 measures: - Patient's assessment of RA pain (visual analogue scale (VAS) 100 mm), -Patient's global assessment of disease activity (VAS 100 mm), -Physician's global assessment of disease activity (VAS 100 mm), -Patient self-assessed disability index(HAQ-DI© score), -Acute phase reactant (CRP or ESR). ACR50 and ACR70 responses were defined as ACR20 response replacing "20% improvement" by "50% improvement" and "70% improvement", respectively.
Time Frame: Week 4, week 12 and week 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 127 | 138
Participants
  ACR20 response Week 4: number analyzed (Participants) | 126 | 138
  ACR20 response Week 4 | 64 | 71
  ACR20 response Week 12 | 100 | 106
  ACR20 response Week 24 | 111 | 130
  ACR50 response Week 4: number analyzed (Participants) | 126 | 138
  ACR50 response Week 4 | 25 | 25
  ACR50 response Week 12 | 53 | 67
  ACR50 response Week 24 | 78 | 98
  ACR70 response Week 4: number analyzed (Participants) | 126 | 138
  ACR70 response Week 4 | 7 | 9
  ACR70 response Week 12 | 24 | 35
  ACR70 response Week 24 | 48 | 53

9. Secondary Outcome: Study Period 1 - Changes From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI©) at Weeks 4, 12 and 24;
Description: Health assessment questionnaire (HAQ-DI) disability index ranges from 0 (best) to 3 (worst).The HAQ© was scored in accordance with the recommendation from the developers outlined in the "HAQ PACK" from Stanford University, California.
  Ramey Dr, Fries JF, Singh G. in B. Spilker Quality of Life and Pharmacoleconomics in Clinical Trials, 2nd ed, The Health Assessment Questionnaire 1995 -- Status and Review. Philadelphia: Lippincott-Raven Pub., 1996, p 227 - 237.
  Fries JF, Spitz P, Kraines G, Holman H. Measurement of Patient Outcome in Arthritis, Arthritis and Rheumatism, 1980, 23:137-145.
Time Frame: Weeks 4, 12 and 24;
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 127 | 138
score on a scale
  Week 4 | -0.32 (0.519) | -0.32 (0.449)
  Week 12 | -0.50 (0.576) | -0.47 (0.501)
  Week 24 | -0.63 (0.610) | -0.59 (0.543)

10. Secondary Outcome: Study Period 1- Proportion of Patients Achieving HAQ-DI© in Normal Range (≤ 0.5) at Weeks 4, 12 and 24;
Description: Health assessment questionnaire disability index (HAQ-DI©) ranges from 0 (best) to 3 (worst)
Time Frame: Weeks 4, 12 and 24;
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 127 | 138
Participants
  Week 4: number analyzed (Participants) | 125 | 138
  Week 4 | 27 | 33
  Week 12 | 38 | 40
  Week 24 | 46 | 50

11. Secondary Outcome: Study Period 1- Proportion of Patients Achieving HAQ-DI© Score Improvement >0.3 at Weeks 4, 12 and 24
Description: Health assessment questionnaire (HAQ-DI©) disability index ranges from 0 (best) to 3 (worst)
Time Frame: Weeks 4, 12 and 24;
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 127 | 138
Participants
  Week 4: number analyzed (Participants) | 125 | 138
  Week 4 | 106 | 117
  Week 12 | 102 | 109
  Week 24 | 91 | 106

12. Secondary Outcome: Study Period 1 - Functional Assessment of Chronic Illness Therapy (FACIT©) Fatigue Scale Relative to Baseline at Weeks 4, 12 and 24 (Change From Baseline)
Description: FACIT© fatigue scale is a 13- item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function, ranging from 0 (worst) to 52 (best).
Time Frame: Weeks 4, 12 and 24;
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 127 | 138
score on a scale
  Week 4 | 6.59 (7.949) | 7.25 (8.591)
  Week 12 | 10.49 (9.218) | 10.62 (9.134)
  Week 24 | 12.57 (10.760) | 12.72 (9.451)

13. Secondary Outcome: Study Period 1 - CRP (C-reactive Protein) Changes From Baseline in GP2017 and US-licensed Humira Treated at Weeks 4, 12 and 24
Description: Outcome measure 13 presents changes in CRP measures in blood while Outome measure 7 presents changes in DAS28-CRP scores (calculated composite score to measure the disease activity)
Time Frame: Week 4, week 12, week 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 127 | 138
mg/L
  CRP change from baseline week 4 | -4.79 (8.728) | -4.93 (12.128)
  CRP change from baseline week 12 | -5.98 (11.270) | -5.07 (11.791)
  CRP change from baseline week 24 | -2.51 (19.176) | -5.30 (13.726)

14. Secondary Outcome: Study Period 1 -ESR (Erythrocyte Sedimentation Rate) Changes From Baseline in GP2017 and US-licensed Humira Treated at Weeks 4, 12 and 24
Description: Outcome measure 13 presents changes in ESR measures in blood while outcome measure 7 presents changes in DAS28-ESR scores (calculated composite score to measure the disease activity)
Time Frame: Week 4, week 12, week 24
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 127 | 138
mm/h
  ESR change from baseline week 4 | -16.17 (14.693) | -13.98 (15.823)
  ESR change from baseline week 12 | -17.33 (16.214) | -15.08 (31.150)
  ESR change from baseline week 24 | -19.60 (20.494) | -20.49 (18.255)

15. Secondary Outcome: Study Period 1: Incidence and Severity of Injection Site Reactions in GP2017 and Humira
Description: Incidence of injection site reactions in GP2017 and Humira
Time Frame: Treatment Period 1, 24 weeks
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 177 | 176
Participants
  incidence of injection site reactions | 7 | 11
  injection site reactions MILD | 7 | 7
  injection site reactions MODERATE | 0 | 4
  injection site reactions SEVERE | 0 | 0
  Injection site erythema | 2 | 6
  Injection site pruritus | 2 | 3
  Injection site pain | 2 | 1
  Injection site inflammation | 2 | 0
  Injection site rash | 0 | 2
  Injection site discolouration | 0 | 1

16. Secondary Outcome: Study Period 1 - Immunogenicity by Measuring the Rate of Anti-drug Antibody (ADA) Formation Against Adalimumab in Patients Treated With GP2017 or Humira (Positive Patients)
Description: Frequency of patients having anti-drug antibody (ADA) during 24 weeks
Time Frame: baseline, week 2, week 4, week 12, week 24
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 177 | 176
Participants
  Baseline: number analyzed (Participants) | 176 | 174
  Baseline | 10 | 6
  Week 2: number analyzed (Participants) | 160 | 166
  Week 2 | 12 | 10
  Week 4: number analyzed (Participants) | 159 | 166
  Week 4 | 14 | 22
  Week 12: number analyzed (Participants) | 157 | 164
  Week 12 | 16 | 23
  Week 24: number analyzed (Participants) | 151 | 162
  Week 24 | 23 | 25

17. Secondary Outcome: Study Period 2 - Immunogenicity by Measuring the Rate of Anti-drug Antibody (ADA) Formation Against Adalimumab in Patients Treated With GP2017 Who Continued GP2017 or Switched to GP2017 From Humira (Positive Patients)
Description: Frequency of patients having anti-drug antibody (ADA) during 24 weeks
Time Frame: week 24, week 36, week 48
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 159 | 166
Participants
  Week 24: number analyzed (Participants) | 148 | 160
  Week 24 | 22 | 25
  Week 36: number analyzed (Participants) | 140 | 153
  Week 36 | 21 | 22
  Week 48: number analyzed (Participants) | 113 | 127
  Week 48 | 12 | 12

18. Secondary Outcome: Study Period 2 : Proportion of Patients Achieving ACR20/50/70 Response at Week 48, in Patients Treated With GP2017 Who Continued GP2017 or Switched to GP2017 From Humira
Time Frame: week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 108 | 126
Participants
  ACR20 response Week 48 | 93 | 111
  ACR50 response Week 48 | 72 | 81
  ACR70 response Week 48 | 49 | 55

19. Secondary Outcome: Study Period 2 - Health Assessment Questionnaire-Disability Index (HAQ-DI©) Changes From Week 24 at Week 48 in Patients Treated Continuously With GP2017 and in Patients Treated With GP2017 After Switch From Humira
Description: Health assessment questionnaire (HAQ-DI) disability index ranges from 0 (best) to 3 (worst)
Time Frame: Weeks 48
Population: Treatment period 1 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 108 | 126
score on a scale | 0.01 (0.358) | -0.03 (0.427)

20. Secondary Outcome: Study Period 2 :Proportion of Patients Treated Continuously With GP2017 and Patients Treated With GP2017 After Switch From Humira Achieving HAQ-DI© Score in Normal Range ≤0.5 at Week 48
Time Frame: week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Count of Participants; unit: Participants
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 108 | 126
Participants | 45 | 52

21. Secondary Outcome: Study Period 2 : Functional Assessment of Chronic Illness Therapy (FACIT©) Fatigue Scale Changes From Week 24 at Week 48 in Patients Treated Continuously With GP2017 and in Patients Treated With GP2017 After Switch From Humira
Description: FACIT©: from 0 (worst) to 52 (best), a score of less than 30 indicates severe fatigue
Time Frame: week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 108 | 126
score on a scale | -0.65 (7.421) | -0.85 (7.476)

22. Secondary Outcome: Study Period 2: Changes From Week 24 at Week 48 in DAS28-CRP and DAS28-ESR Scores in Patients Treated Continuously With GP2017 and in Patients Treated With GP2017 After Switch From Humira
Description: DAS28-CRP is a disease activity score and defined in primary outcome measure. DAS28-ESR is the DAS28 erythrocyte sedimentation rate score.
  DAS28-CRP and DAS28-ESR:
  1. best is 0,
  2. < 2.6 - remission,
  3. ≥ 2.6 to ≤ 3.2 - low disease activity
  4. > 3.2 to ≤ 5.1 - moderate disease activity
  5. > 5.1 - high disease activity
  DAS28-ESR = 0.56 * sqrt(tender28) + 0.28* sqrt(swollen28) + 0.7 * ln(ESR) + 0.014 * GDA where • tender28 and swollen28 are the number of tender and swollen joints as assessed using 28-joint count • CRP is C-reactive protein (mg/l) • ESR is erythrocyte sedimentation rate (mm/h) • GDA is the global disease activity measured on a Visual Analogue Scale (VAS) of 100 mm.Values range from 0 to 10. Higher values mean a higher disease activity.
Time Frame: week 48
Population: Treatment period 2 per protocol set. Patients with data available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 108 | 126
score on a scale
  DAS28-CRP Week 48, change from week 24: number analyzed (Participants) | 107 | 125
  DAS28-CRP Week 48, change from week 24 | -0.10 (0.893) | 0.00 (0.941)
  DAS28-ESR Week 48, change from week 24 | -0.04 (1.015) | 0.00 (1.025)

23. Secondary Outcome: Study Period 2: Incidence of Injection Site Reactions in Patients Treated Continuously With GP2017 and in Patients Treated With GP2017 After Switch From Humira
Description: Incidence of injection site reactions
Time Frame: up to 48 weeks
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2017 | Humira / Switched GP2017
Number analyzed (Participants) | 159 | 166
Participants
  Number of patients with ISRs | 1 | 2
  Injection site erythema | 1 | 2
  Injection site pruritus | 0 | 1
  injection site reactions MILD | 1 | 1
  injection site reactions MODERATE | 0 | 1
  injection site reactions SEVERE | 0 | 0

ADVERSE EVENTS:
Time Frame: Each patient was followed up for safety during the whole study treatment duration ( approximately 24 months) , and Adverse Events were collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) for every single patient, + 30 day safety follow up period after study treatment discontinuation.
Description: AE additional description
Groups:
- Study Period 1 SP1 SAF GP2017: Study Period 1 SP1 SAF GP2017
- Study Period 1 SP1 SAF Humira: Study Period 1 SP1 SAF Humira
- Study Period 2 SP2 SAF Continued GP2017: Study Period 2 SP2 SAF Continued GP2017
- Study Period 2 SP2 SAF Humira to GP2017: Study Period 2 SP2 SAF Humira to GP2017
- Entire Study SP1 SAF GP2017: Entire study SP1 SAF GP2017
- Entire Study SP1 SAF Humira/Switched GP2017: Entire study SP1 SAF Humira/Switched GP2017
Arm/Group | Study Period 1 SP1 SAF GP2017 | Study Period 1 SP1 SAF Humira | Study Period 2 SP2 SAF Continued GP2017 | Study Period 2 SP2 SAF Humira to GP2017 | Entire Study SP1 SAF GP2017 | Entire Study SP1 SAF Humira/Switched GP2017
All-Cause Mortality (participants affected / at risk) | 0/177 | 0/176 | 0/159 | 0/166 | 0/177 | 0/176
Serious Adverse Events (participants affected / at risk) | 5/177 | 4/176 | 4/159 | 6/166 | 7/177 | 10/176
Other Adverse Events (participants affected / at risk) | 83/177 | 74/176 | 28/159 | 26/166 | 94/177 | 80/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Period 1 SP1 SAF GP2017 (N=177) | Study Period 1 SP1 SAF Humira (N=176) | Study Period 2 SP2 SAF Continued GP2017 (N=159) | Study Period 2 SP2 SAF Humira to GP2017 (N=166) | Entire Study SP1 SAF GP2017 (N=177) | Entire Study SP1 SAF Humira/Switched GP2017 (N=176)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hemianopia homonymous (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Study Period 1 SP1 SAF GP2017 (N=177) | Study Period 1 SP1 SAF Humira (N=176) | Study Period 2 SP2 SAF Continued GP2017 (N=159) | Study Period 2 SP2 SAF Humira to GP2017 (N=166) | Entire Study SP1 SAF GP2017 (N=177) | Entire Study SP1 SAF Humira/Switched GP2017 (N=176)
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 2 | 0 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 7 | 0 | 0 | 4 | 7
Nausea (Gastrointestinal disorders) | 5 | 1 | 0 | 0 | 5 | 1
Fatigue (General disorders) | 5 | 0 | 0 | 1 | 5 | 1
Injection site erythema (General disorders) | 2 | 6 | 1 | 2 | 3 | 6
Bronchitis (Infections and infestations) | 4 | 8 | 1 | 4 | 4 | 12
Gastroenteritis (Infections and infestations) | 2 | 4 | 1 | 0 | 3 | 4
Influenza (Infections and infestations) | 3 | 5 | 1 | 0 | 4 | 5
Oral herpes (Infections and infestations) | 4 | 3 | 1 | 0 | 5 | 3
Pharyngitis (Infections and infestations) | 9 | 10 | 1 | 3 | 10 | 10
Sinusitis (Infections and infestations) | 5 | 3 | 0 | 2 | 5 | 5
Upper respiratory tract infection (Infections and infestations) | 12 | 7 | 4 | 3 | 14 | 9
Urinary tract infection (Infections and infestations) | 4 | 6 | 2 | 3 | 6 | 8
Viral upper respiratory tract infection (Infections and infestations) | 26 | 16 | 4 | 4 | 29 | 19
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 1 | 2 | 4
Transaminases increased (Investigations) | 0 | 3 | 1 | 1 | 1 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 3 | 2 | 0 | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 0 | 2 | 0 | 10 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5 | 2 | 6 | 3
Headache (Nervous system disorders) | 7 | 5 | 2 | 2 | 8 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0 | 5 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1 | 0 | 4
Hypertension (Vascular disorders) | 5 | 3 | 2 | 1 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT02744755/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT02744755/SAP_001.pdf